CLINICAL TRIAL: NCT03191552
Title: The Effect of Vest Type Dynamic Elastomeric Fabric Orthosis (DEFO) on Sitting Balance and Gross Manuel Dexterity in Children With Bilateral Cerebral Palsy: A Feasibility and Randomized, Single-blinded, Pilot Study
Brief Title: The Effect of Dynamic Elastomeric Fabric Orthosis (DEFO) on Sitting Balance and Gross Manuel Dexterity in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2013.0351
Record Dates: First submitted 2017-06-08; First posted 2017-06-19 (Actual); Results first posted 2017-12-14 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Cerebral Palsy; Postural; Defect
Keywords: Cerebral palsy; lycra garments; orthosis; suit therapy; trunk control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Observational Model: Cohort Time Perspective: Prospective Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPIO 2 hours (Experimental): All children will be hospitalized for 2 weeks and will receive conventional exercise therapy including range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills during hospital inpatient stay throughout 2 weeks 2 hours a day.
  SPIO 2 hours group will receive conventional exercise therapy with the garment on for 2 hours.
  Interventions: Device: SPIO; Other: conventional exercises
- SPIO 6 hours (Experimental): SPIO 6 hours group will receive conventional exercise therapy with the garment on for 2 hours and worn SPIO 4 hours more in addition to 2 hour of wear during exercise therapy.
  Interventions: Device: SPIO; Other: conventional exercises
- Control(conventional exercises) (Active Comparator): Control group will only receive conventional exercise therapy (for two hours a day) including range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills during hospital inpatient stay throughout 2 weeks
  Interventions: Other: conventional exercises

INTERVENTIONS:
Device: SPIO — SPIO (stabilizing input pressure orthosis) 2 hours will receive conventional exercise therapy with the garment on during 2 hours. SPIO 6 hours group wore the SPIO 4 hours more in addition to 2 hours during therapy.
  SPIO 6 hours group will wear the SPIO 4 hours more in addition to 2 hours during therapy.
  (conventional exercises :range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills
  Arms: SPIO 2 hours; SPIO 6 hours
Other: conventional exercises — range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills

SUMMARY:
To evaluate the effects and feasibility of lycra based compression garment called Stabilizing Pressure Input Orthosis (SPIO) vest on posture and balance during sitting and gross manuel dexterity, parent satisfaction with the garment and to to compare 2 hours vs 6 hours of daily wear time.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a disorder of development of movement and posture due to non-progressive lesion in fetal or infant brain. Postural control in children with cerebral palsy (CP) is deteriorated due to inappropriate muscle force and lack of sensory integration. The trunk which is found in the centre of the body plays a crucial role in postural control. Research and treatments in CP have focused on extremities rather than trunk control. Both evaluation and treatment of trunk impairment have not been adequately addressed in previously published studies. Improved proximal stability obtained by a better trunk control may lead to improvements in upper extremity function.

Dynamic elastomeric fabric orthosis (DEFO) which are lycra based compression garments provide extra proprioceptive information which enhances body awareness. The more correct proprioceptive input result in the more proper alignment. Vest type dynamic elastomeric fabric orthosis (DEFO) is composed of a front part which is compromised of double-or triple-layer of lycra fabric attached to velcro sensitive neoprene back panel. Thus, it provides adjustable compression around the shoulder, trunk, pelvis, and hips. It is proposed that these orthotic garments provides stabilization of the trunk, shoulder and pelvis girdle and thus improve proximal stability and upper extremity function. Children with sensory deficits and poor muscle strength including children with neuromotor developmental disorders and hypotonia can benefit from the use of vest type dynamic elastomeric fabric orthosis. Severe restricted pulmonary function and refractory cyanosis are absolute contraindications for lycra based orthosis use while having severe reflux symptoms, uncontrolled epilepsy, cardiovascular circulatory disorders and being diagnosed with diabetes are relative contraindications. The adverse events pertaining to the use of these orthoses are difficulty in donning/doffing, toileting problems such as constipation and urinary leakage, decrease in respiratory function, heat and skin discomfort. Due to those unwanted effects, it can be assumed that longer wear time of the orthosis may lower compliance. However, the optimal wear time for vest type dynamic elastomeric fabric orthosis has not been established so far. The reported wear time of suit therapies range from 2 to12 hours a day during 2-12 weeks. The aim of this study was to investigate if the use of a vest type dynamic elastomeric fabric orthosis (DEFO) vest type dynamic elastomeric fabric orthosis is feasible or not and will lead to improvement in sitting balance, sitting as a gross motor function and gross manuel dexterity. The secondary purposes of the present study are to evaluate parent satisfaction with the orthosis and to compare 2 hours vs 6 hours of daily wear time.

ELIGIBILITY:
Inclusion Criteria:

1. being classified at Gross Motor Function Classification System (GMFCS) level III-IV
2. being classified at Manual Ability Classification System (MACS) level III-IV
3. being able to understand and execute given instructions for evaluations
4. parental acceptance of using the lycra based compression garment.

Exclusion Criteria:

1. serious respiratory restriction
2. having refractory cyanosis or circulatory disorder
3. having undergone lycra compression orthosis treatment programme previously
4. having undergone botulinum toxin injection within last 3 months or orthopedic surgery within 1 year
5. severe scoliosis (Cobb angle (CA) >40°)
6. uncontrolled epilepsy
7. having intrathecal baclofen pump
8. having undergone selective dorsal rhizotomy
9. having reflux more than 3 times a week.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esra Giray, MD, Principal Investigator — Marmara University School of Medicine, Department of Physical Medicine and Rehabilitation; Naime Evrim Karadag-Saygi, Prof, Study Chair — Marmara University School of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blair E, Ballantyne J, Horsman S, Chauvel P. A study of a dynamic proximal stability splint in the management of children with cerebral palsy. Dev Med Child Neurol. 1995 Jun;37(6):544-54. doi: 10.1111/j.1469-8749.1995.tb12041.x. PMID 7789663
- [Result] How does the TherSuit® works? TheraSuit® / TheraSuit Method®. http://www.suittherapy.com/therasuit%20info.htm.
- [Result] Hylton N, Schoos KK. Deep Pressure Sensory Input. SPIO Flexible Compression Bracing. http://www.spioworks.com/files/Deep%20Pressure%20Sensory%20Input%20Hylton%20Schoos.pdf; 2007.
- [Result] Christy JB, Steed L. Commentary on "The effect of suit wear during an intensive therapy program in children with cerebral palsy". Pediatr Phys Ther. 2011 Summer;23(2):143. doi: 10.1097/PEP.0b013e318219352d. No abstract available. PMID 21552074
- [Result] Hylton N, Allen C. The development and use of SPIO Lycra compression bracing in children with neuromotor deficits. Pediatr Rehabil. 1997 Apr-Jun;1(2):109-16. doi: 10.3109/17518429709025853. PMID 9689245
- [Result] Knox V. The use of Lycra garments in children with cerebral palsy: A report of a descriptive clinical trial. The British Journal of Occupational Therapy 2003; 66: 71-7.
- [Result] Matthews M, Crawford R. The use of dynamic Lycra orthosis in the treatment of scoliosis: a case study. Prosthet Orthot Int. 2006 Aug;30(2):174-81. doi: 10.1080/03093640600794668. PMID 16990228
- [Result] Saavedra S. Trunk control in cerebral palsy: are we ready to address the elephant in the room? Dev Med Child Neurol. 2015 Apr;57(4):309-10. doi: 10.1111/dmcn.12614. Epub 2014 Nov 20. No abstract available. PMID 25412796
- [Result] Myhr U, von Wendt L. Improvement of functional sitting position for children with cerebral palsy. Dev Med Child Neurol. 1991 Mar;33(3):246-56. doi: 10.1111/j.1469-8749.1991.tb05114.x. PMID 1760002
- [Result] Myhr U, von Wendt L, Norrlin S, Radell U. Five-year follow-up of functional sitting position in children with cerebral palsy. Dev Med Child Neurol. 1995 Jul;37(7):587-96. doi: 10.1111/j.1469-8749.1995.tb12047.x. PMID 7615145
- [Derived] Giray E, Karadag-Saygi E, Ozsoy T, Gungor S, Kayhan O. The effects of vest type dynamic elastomeric fabric orthosis on sitting balance and gross manual dexterity in children with cerebral palsy: a single-blinded randomised controlled study. Disabil Rehabil. 2020 Feb;42(3):410-418. doi: 10.1080/09638288.2018.1501098. Epub 2018 Oct 7. PMID 30293457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 36 children evaluated for recruitment, 26 of them met the inclusion criteria. There were two drop-outs throughout the follow-up period. Finally, data from 24 children were analyzed.
Pre-assignment Details: Not meeting inclusion criteria (n=10)
  * Mixed CP n=2
  * Undergone surgery in past 6 months n=2
  * BTX-A injection in past 3 months n=2
  * Who do not understand and execute given instructions, severe CP n=4
Groups:
- SPIO(Stabilizing Pressure Input Orthosis) 2 Hours: All children will be hospitalized for 2 weeks and will receive conventional exercise therapy including range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills during hospital inpatient stay throughout 2 weeks 2 hours a day.
  SPIO 2 hours group will receive conventional exercise therapy with the garment on for 2 hours.
  SPIO (stabilizing input pressure orthosis): SPIO 2 hours will receive conventional exercise therapy with the garment on during 2 hours. SPIO 6 hours group wore the SPIO 4 hours more in addition to 2 hours during therapy.
  SPIO 6 hours group will wear the SPIO 4 hours more in addition to 2 hours during therapy.
  (conventional exercises :range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills
  conventional exercises: range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross
- SPIO (Stabilizing Pressure Input Orthosis) 6 Hours: SPIO 6 hours group will receive conventional exercise therapy with the garment on for 2 hours and worn SPIO 4 hours more in addition to 2 hour of wear during exercise therapy.
  SPIO (stabilizing input pressure orthosis): SPIO 2 hours will receive conventional exercise therapy with the garment on during 2 hours. SPIO 6 hours group wore the SPIO 4 hours more in addition to 2 hours during therapy.
  SPIO 6 hours group will wear the SPIO 4 hours more in addition to 2 hours during therapy.
  (conventional exercises :range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills
  conventional exercises: range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills
- Control (Conventional Exercises): Control group will only receive conventional exercise therapy (for two hours a day) including range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills during hospital inpatient stay throughout 2 weeks
  conventional exercises: range of motion, strengthening, trunk control and strengthening exercises and exercises to improve fine and gross motor skills
Period: Overall Study
Arm/Group | SPIO(Stabilizing Pressure Input Orthosis) 2 Hours | SPIO (Stabilizing Pressure Input Orthosis) 6 Hours | Control (Conventional Exercises)
Started | 9 | 9 | 8
Completed | 8 | 8 | 8
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Undergone surgery (Progressive hip dyspl | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SPIO 2 Hours: SPIO 2 hours (worn SPIO 2 hours during therapy)
  9 were allocated, one of them lost follow up before the assessment at 1 month and 8 completed
- SPIO 6 Hours: SPIO 6 hours (worn SPIO 4 hours in addition to 2 hours of wear during therapy).
  9 were allocated, one of them withdrew due to surgery for progressive hip dysplasia between the assessments at 1 month and 3 months and 8 completed.
- Control (Conventional Exercises): Control group (received only conventional exercise therapy) 8 were recruited/ 8 completed the study
- Total: Total of all reporting groups
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 8 | 24
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 64.29 (18.09) | 60.5 (19.57) | 55.63 (18.11) | 61 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 6 | 7 | 6 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cerebral palsy (CP) type [Count of Participants; unit: Participants]
  Diplegic | 1 | 0 | 1 | 2
  Tetraplegic | 7 | 8 | 7 | 22
GMFCS Level [Count of Participants; unit: Participants] — GMFCS© Robert Palisano, Peter Rosenbaum, Stephen Walter, Dianne Russell, Ellen Wood, Barbara Galuppi, 1997. CanChild Centre for Childhood Disability Research, McMaster University. (Reference: Dev Med Child Neurol 1997;39:214-223).
  Levels I-V based on self-initiated movement, with emphasis on sitting, transfers, and mobility. Level I is highest functioning, level V is lowest
  General:
  I: walks without limitations II: walks with limitations III: walks using hand-held mobility device IV: self-mobility with limitations; may use powered mobility V: transported in manual wheelchair
  Participants
    GMFCS level 3 | 2 | 2 | 1 | 5
    GMFCS level 4 | 6 | 6 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Sitting Assessment Scale
Description: Sitting Assessment Scale was devoloped for observational assessment of posture and balance during sitting after seating interventions. The scale consists of 5 items including head control, trunk control, foot control, arm function and hand function which are assessed as follows: 1= none; 2= poor; 3= fair; 4= good). The minimum and maximum possible scores are 5 to 20 respectively.
Time Frame: Immediate after orthosis is worn
Population: The immediate effect of orthosis could only be evaluated in SPIO groups because the orthosis is tailor made and only children in SPIO groups had the orthosis. Given that the number of the objects in each SPIO group is 8, immediate effect of the orthosis could only be evaluated in children recruited in SPIO groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Before Treatment: SPIO groups before treatment (orthosis is tailor made and only children in SPIO groups had the orthosis so the arm control (conventinal exercises) group is not included)
- Immediately After Orthosis Worn: Immediate evaluation after orthosis worn
Arm/Group | Before Treatment | Immediately After Orthosis Worn
Number analyzed (Participants) | 16 | 16
units on a scale | 12.56 (2.4) | 15.06 (2.54)
Statistical Analysis 1: Comparison: Before Treatment; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Sitting Assessment Scale
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SPIO 2 Hours: SPIO 2 hours (worn SPIO 2 hours during therapy)
- SPIO 6 Hours: SPIO 6 hours (worn SPIO 4 hours in addition to 2 hours of wear during therapy)
- Control (Conventional Exercises): Control group (received only conventional exercise therapy),
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 16.8 (3.15) | 18 (1.7) | 14.8 (2.6)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.027, Kruskal-Wallis — Mann-Whitney U test was used to test the significance of pairwise differences using Bonferroni correction to adjust for multiple comparisons.p value of less than 0.05/3 was determined as the level of statistical significance

3. Primary Outcome: Sitting Assessment Scale
Description: as for outcome 1
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 17.5 (2.27) | 18.63 (1.85) | 15.13 (1.1)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.008, Kruskal-Wallis — Mann-WhitneyU test was used to test the significance of pairwise differences using Bonferroni correction to adjust for multiple comparisons.p value of less than 0.05/3 was determined as the level of statistical significance

4. Primary Outcome: Sitting Assessment Scale
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 17.75 (1.75) | 19.38 (1.19) | 1.63 (2.33)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority — Mann-WhitneyU test was used to test the significance of pairwise differences using Bonferroni correction to adjust for multiple comparisons.p value of less than 0.05/3 was determined as the level of statistical significance; p = 0.004, Kruskal-Wallis — Mann-WhitneyU test was performed to test the significance of pairwise differences using Bonferroni correction to adjust for multiple comparisons.p value of less than 0.05/3 was determined as the level of statistical significance

5. Secondary Outcome: Gross Motor Function Measure-B, Sitting Dimension
Description: Evaluates degree of achievement of sitting as a gross motor function. Gross Motor Function Measure sitting dimension is composed of 20 items. Each tem is scored according to special instructions on GMFM Manuel with a 4-point Likert scale including 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. If it is not possible to test an item, it should be noted as not tested (NT) It assesses degree of achievement of gross motor functions rather than quality of them. Minimum score is 0 while maxium score is 60(3x20).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 36.88 (14.16) | 37 (11.26) | 34 (7.69)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.837, Kruskal-Wallis

6. Secondary Outcome: Gross Motor Function Measure-B, Sitting Dimension
Description: as for outcome 5
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 43.25 (12.24) | 40.88 (11.68) | 37.25 (9.68)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.570, Kruskal-Wallis

7. Secondary Outcome: Gross Motor Function Measure-B, Sitting Dimension
Description: as for outcome 5
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 45 (9.04) | 45.38 (7.52) | 39.25 (10.3)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.334, Kruskal-Wallis

8. Secondary Outcome: Box and Block Test (BBT)
Description: Evaluates gross manuel dexterity. Box and Block Test which consists of a box divided into two compartments by a partition and blocks with standardized dimensions is used to assess unilateral gross manuel dexterity. The object is instructed to transport boxes one by one from one compertmant of the box to other in 60 seconds. The object should sit on a chair with a standard height and face the box. He/she should practice for a 15 second trial period before testing. If two blocks are carried at the same time, it is counted as one. And also if the block falls on the floor after it has been carried across, it is still counted. The score is the number of boxes transferred from one compartment to other in 60 seconds.
Time Frame: Immediate after orthosis is worn
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Before Treatment: Box and Block Test Score of SPIO groups before Treatment (orthosis is tailor made and only children in SPIO groups had the orthosis so the arm control (conventinal exercises) group is not included)
- İmmediate After Orthosis Wear: Box and Block Test Score of SPIO groups immediate after the orthosis wear (orthosis is tailor made and only children in SPIO groups had the orthosis so the arm control (conventinal exercises) group is not included)
Arm/Group | Before Treatment | İmmediate After Orthosis Wear
Number analyzed (Participants) | 16 | 16
units on a scale | 10.18 (4.35) | 15.06 (2.54)
Statistical Analysis 1: Comparison: Before Treatment vs İmmediate After Orthosis Wear; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Box and Block Test (BBT)
Description: as for outcome 8
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 14 (7.27) | 12.63 (4.93) | 14.75 (5.73)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.77, Kruskal-Wallis

10. Secondary Outcome: Box and Block Test (BBT)
Description: as for outcome 8
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 14.75 (6.76) | 14 (5.4) | 15.5 (6.21)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.889, Kruskal-Wallis

11. Secondary Outcome: Box and Block Test (BBT)
Description: as for outcome 8
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 15.63 (8.23) | 14.88 (3.91) | 15.75 (5.99)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.956, Kruskal-Wallis

12. Secondary Outcome: Parent Satisfaction Questionnaire (Sum of the Items 3,5 and 7)
Description: A non-standardised 5-point Likert type scale was invented by the investigators to assess compliance and satisfaction with wearing orthosis. The parent satisfaction survey was measured on a 5-point Likert scale with 1 strongly agree and 5 strongly disagree to items of questionnaire below:
  Parent satisfaction survey
  1. SPIO vest was easy to put on/off.
  2. Child was comfartable during times the SPIO was worn.
  3. Child's sitting balance improved.
  4. Caring of the garment (cleaning vs) was easy.
  5. Child's confidence was improved.
  6. No problems about touletting occured.
  7. I wish to attend this therapy programme again.
  8. I consider attending this therapy programme in the future again.
  9. I consider to use SPIO vest for my child after the the therapy programme ended. Higher values representing better outcome. Items 3,5 and 7 is used to compare all groups (min 3-max 15) while the all of the items were used to compare the SPIO 2 hours and SPIO 6 hours (min 5-max 45).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 11.43 (0.97) | 11.5 (0.76) | 8.5 (2.27)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0,001, Kruskal-Wallis — [p-value comment as in outcome 3, analysis 1]

13. Secondary Outcome: Parent Satisfaction Questionnaire (Sum of the Items 3,5 and 7)
Description: as for outcome 12
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 11.43 (0.79) | 11 (0.93) | 9 (3.3)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.14, Kruskal-Wallis

14. Secondary Outcome: Parent Satisfaction Questionnaire (Sum of the Items 3,5 and 7)
Description: as for outcome 12
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale | 11.14 (1.07) | 11 (0.93) | 9.25 (2.05)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours vs Control (Conventional Exercises); Test type: Superiority; p = 0.08, Kruskal-Wallis

15. Secondary Outcome: Parent Satisfaction Questionnaire Total Score
Description: as for outcome 12
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours
Number analyzed (Participants) | 8 | 8
units on a scale | 31.14 (1.07) | 30.13 (2.59)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours; Test type: Superiority; p = 0.314, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Parent Satisfaction Questionnaire Total Score
Description: as for outcome 12
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours
Number analyzed (Participants) | 8 | 8
units on a scale | 31.14 (1.21) | 30.63 (1.3)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours; Test type: Superiority; p = 0.244, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Parent Satisfaction Questionnaire Total Score
Description: as for outcome 12
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIO 2 Hours | SPIO 6 Hours
Number analyzed (Participants) | 8 | 8
units on a scale | 31.29 (1.11) | 30 (2.33)
Statistical Analysis 1: Comparison: SPIO 2 Hours vs SPIO 6 Hours; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SPIO 2 Hours | SPIO 6 Hours | Control (Conventional Exercises)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Outcome measures assesses body structure and function only. Effects of orthosis on activity and participation were not evaluated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03191552/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03191552/SAP_001.pdf
  • Informed Consent Form (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03191552/ICF_002.pdf